CLINICAL TRIAL: NCT01840384
Title: Longitudinal Study on the Effect of Multiple Micro Nutrients Supplementation on Haemoglobin Level of 8 to 22-month-old Indonesian Children.
Brief Title: Efficacy Study of Multiple Micro Nutrients Supplementation
Acronym: Babytop
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PT. Sari Husada (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CT.01.2012
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Anemia, Iron-deficiency
Keywords: Healthy infants; Anemia, iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — maltodextrin; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-micronutrients (Experimental): Multi-micronutrients
  Interventions: Dietary Supplement: Multi-micronutrients
- Maltodextrin and Lactose (Placebo Comparator): Placebo contained maltodextrin and lactose
  Interventions: Dietary Supplement: Maltodextrin and Lactose

INTERVENTIONS:
Dietary Supplement: Multi-micronutrients
  Arms: Multi-micronutrients
Dietary Supplement: Maltodextrin and Lactose
  Arms: Maltodextrin and Lactose

SUMMARY:
This study is initiated to investigate the effect of multi micronutrient supplementation for 12 months on serum haemoglobin level in Indonesian young children.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy Indonesian infants
* Age 8-10 month at baseline visit
* Willing to take 2 sachets of study product per day
* Planning to reside in the study area during the next 14-16 months
* Written informed consent by parent(s) or legally acceptable representative (in ICF there is statement that both are agree that child participate in the study)

Exclusion Criteria:

* Haemoglobin < 8 g/dL at screening visit*.
* Significant congenital abnormality which according to investigator's clinical judgement will interfere the study conduct and assessment
* Any known conditions likely to affect nutrient absorption diagnosed by the child's physician
* Disorders requiring a special diet (such as food intolerance or food allergy or complaints such as reflux, constipation and cramps for which special formula is required).
* Any other current or previous illnesses/conditions or intervention which according to investigator's clinical judgement could interfere the study conduct and assessment (e.g. chronic illness or physical or mental handicaps)
* Regular use of MMN supplements syrup (every day in > 1 week) within two weeks prior to entry into the study.
* Not intending to use micronutrient supplements during the study
* Participation in any other studies involving similar investigational or marketed products concomitantly or within two weeks prior to entry into the study.
* Premature birth (gestational age <37 weeks)
* Low birth weight (< 2500 g)
* Severely under nutrition indicated by any of the following criteria: severely stunted: HAZ < -3 SD; severely underweight WAZ <-3 SD; wasted: WHZ <-2 SD

  *Subject with haemoglobin level (finger prick blood sample) at screening visit between 8-10 g/dL will be given iron syrup supplementation for 1 month. Thereafter, haemoglobin level (whole blood sample) will be checked at baseline visit:
* If Hb > 10 g/dL, subject is eligible for randomisation
* If Hb < 10 g/dL, subject is not eligible for randomisation and will be given iron syrup supplementation for 2 months

Ages: 8 Months to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 239 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Haemoglobin level | 12 months
  Change in serum haemoglobin level after 12 months of intervention

SECONDARY OUTCOMES:
Anemia prevalence | 12 months
  Change in anemia prevalence from baseline to after 12 months of intervention
Anthropometric | 24 months of age
  Change in anthropometric measurements from baseline until 24 months of age
Micronutrients | 12 months
  Change in selected micronutrients status from baseline to after 12 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rini Sekartini, MD, PhD, Principal Investigator — Medical Research Unit, Faculty of Medicine, University of Indonesia
Locations (1):
- Jakarta, Indonesia